CLINICAL TRIAL: NCT04405245
Title: Phase 2 Multi-Center, Double-Masked, Randomized, 28-Day Study to Assess the Efficacy, Safety and Tolerability of Single or Twice Daily Doses of AKB-9778 Ophthalmic Solution as an Adjunct to Latanoprost in Patients With Ocular Hypertension (OHT) or Open Angle Glaucoma (OAG)
Brief Title: Study to Assess the Efficacy, Safety and Tolerability of AKB-9778 Ophthalmic Solution as and Adjunct to Latanoprost in Patients With Ocular Hypertension or Open Angle Glaucoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EyePoint Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AKB-9778-CI-OS-2001
Record Dates: First submitted 2020-05-23; First posted 2020-05-28 (Actual); Results first posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Ocular Hypertension; Primary Open Angle Glaucoma
MeSH Terms: conditions — Ocular Hypertension; Glaucoma, Open-Angle

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- AKB-9778 4% QD + Latanoprost (Experimental): • AKB-9778 4% daily (AM) and placebo for ophthalmic solution daily (PM) plus latanoprost daily (PM) for 28 days
  Interventions: Drug: Latanoprost ophthalmic solution; Drug: AKB-9778 4%
- AKB-9778 4% BID + Latanoprost (Experimental): • AKB-9778 4% twice daily (AM & PM) plus latanoprost daily (PM) for 28 days
  Interventions: Drug: Latanoprost ophthalmic solution; Drug: AKB-9778 4%
- Placebo Twice Daily + Latanoprost (Placebo Comparator): • Placebo for AKB-9778 4% ophthalmic solution twice daily (AM & PM) plus latanoprost daily (PM) for 28 days
  Interventions: Drug: Latanoprost ophthalmic solution; Drug: Placebo

INTERVENTIONS:
Drug: Latanoprost ophthalmic solution — Latanoprost opthalmic solution to be dosed once daily
Drug: AKB-9778 4% — Razuprotafib opthalmic solution
  Arms: AKB-9778 4% BID + Latanoprost; AKB-9778 4% QD + Latanoprost
Drug: Placebo — placebo for razuprotafib opthalmic solution
  Arms: Placebo Twice Daily + Latanoprost

SUMMARY:
This is a phase 2, double masked, randomized, multi-center, parallel-group, 28-day study assessing the safety, tolerability and ocular hypotensive efficacy of AKB-9778 Ophthalmic Solution 4.0% administered once (AM) or twice (AM & PM) daily when used as an adjunctive therapy to latanoprost ophthalmic solution 0.005% once daily (PM) in subjects with elevated IOP due to OAG or OHT.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of OAG or OHT in each eye (OAG in one eye and OHT in the fellow eye is acceptable)
* Must be receiving treatment with a stable regimen of topical prostaglandin eyedrop for a minimum of 2 weeks prior to the Screening Visit; may be taking one additional IOP lowering eyedrop
* IOP of ≥ 18 mmHg and ≤ 27 mmHg in one eye or both eyes at Screening visit
* Following 4 week washout period, IOP ≥ 24 mmHg and < 36 mmHg at 08:00 hour and IOP ≥ 22 mmHg and < 36 mmHg in both eyes at 10:00, 12:00 and 16:00 hours.

Key Exclusion Criteria:

* Clinically significant ocular disease which might interfere with interpretation of the study efficacy endpoints or with safety assessments
* Pseudoexfoliation or pigment dispersion component glaucoma
* History of angle closure glaucoma, or narrow angles or with evidence of peripheral anterior synechiae (PAS) ≥ 180 degrees by gonioscopy within 6 months prior to Screening
* Intraocular pressure ≥ 36 mmHg
* Cup/disc ratio of > 0.8 in either eye
* Severe visual field defect or significant defect (sensitivity of ≤ 10dB) within 10 degrees of fixation in either eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2020-06-06 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2020-11-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - United Medical Research Institute, Inglewood, California
  - North Valley Eye Medical Group, Mission Hills, California
  - Eye Research Foundation, Newport Beach, California
  - North Bay Eye Associates, Petaluma, California
  - Shettle Eye Research, Largo, Florida
  - Clayton Eye Clinical Research, LLC, Morrow, Georgia
  - Coastal Research Associates, Roswell, Georgia
  - Kannarr Eye Care, Pittsburg, Kansas
  - Heart of America Eye Care, P.A., Shawnee Mission, Kansas
  - Tekwani Vision Center, St Louis, Missouri
  - North Valley Eye Medical Group, Rochester, New York
  - Charlotte Eye, Ear, Nose & Throat Assoc. (CEENTA), Charlotte, North Carolina
  - James D. Branch, MD Ophthalmology, Winston-Salem, North Carolina
  - Apex Eye, Cincinnati, Ohio
  - Abrams Eye Center, Cleveland, Ohio
  - Mark J. Weiss, MD, Inc., Tulsa, Oklahoma
  - Scott & Christie and Assoc, Cranberry Township, Pennsylvania
  - Eye Care Specialists, Kingston, Pennsylvania
  - Total Eye Care, Memphis, Tennessee
  - Advancing Vision Research, Nashville, Tennessee
  - Texan Eye / Keystone Research, Austin, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- AKB-9778 4% QD + Latanoprost: • AKB-9778 4% QD (AM) and placebo for AKB-9778 ophthalmic solution QD (PM) plus latanoprost QD (PM) for 28 days
  Latanoprost ophthalmic solution: Latanoprost ophthalmic solution to be dosed once daily
  AKB-9778: AKB-9778 4% ophthalmic solution
- AKB-9778 4% BID + Latanoprost: • AKB-9778 4% BID (AM & PM) plus latanoprost QD (PM) for 28 days
  Latanoprost ophthalmic solution: Latanoprost ophthalmic solution to be dosed once daily
  AKB-9778: AKB-9778 4% ophthalmic solution
- Placebo BID + Latanoprost: • Placebo for AKB-9778 4% ophthalmic solution BID (AM & PM) plus latanoprost QD (PM) for 28 days
  Latanoprost ophthalmic solution: Latanoprost ophthalmic solution to be dosed once daily
  Placebo: placebo for AKB-9778 4% ophthalmic solution
Period: Overall Study
Arm/Group | AKB-9778 4% QD + Latanoprost | AKB-9778 4% BID + Latanoprost | Placebo BID + Latanoprost
Started | 65 | 65 | 64
Completed | 65 | 64 | 64
Not Completed | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Each Baseline participant contributed one study eye and one fellow eye
Units Other Than Participants: Eyes
Groups:
- AKB-9778 4% QD + Latanoprost: • AKB-9778 4%(AM) and placebo for AKB-9778 4% ophthalmic solution daily (PM) plus latanoprost daily (PM) for 28 days
  Latanoprost ophthalmic solution: Latanoprost opthalmic solution to be dosed once daily
  Razuprotafib: razuprotafib opthalmic solution
- AKB-9778 4% BID + Latanoprost: • AKB-9778 4% BID (AM & PM) plus latanoprost daily (PM) for 28 days
  Latanoprost ophthalmic solution: Latanoprost opthalmic solution to be dosed once daily
  Razuprotafib: razuprotafib opthalmic solution
- Placebo Twice Daily + Latanoprost: • Placebo for AKB-9778 4% twice daily (AM & PM) plus latanoprost daily (PM) for 28 days
  Latanoprost ophthalmic solution: Latanoprost opthalmic solution to be dosed once daily
  Placebo: placebo for razuprotafib opthalmic solution
- Total: Total of all reporting groups
Arm/Group | AKB-9778 4% QD + Latanoprost | AKB-9778 4% BID + Latanoprost | Placebo Twice Daily + Latanoprost | Total
Number analyzed (Participants) | 65 | 65 | 64 | 194
Number analyzed (Eyes) | 130 | 130 | 128 | 388
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.3 (8.81) | 65.6 (10.85) | 65.9 (10.55) | 66.6 (10.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 37 | 43 | 120
  Male | 25 | 28 | 21 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 6 | 3 | 18
  Not Hispanic or Latino | 56 | 59 | 61 | 176
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 20 | 17 | 16 | 53
  White | 45 | 47 | 47 | 139
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Diagnosis [Count of Units; unit: Eyes] — Study Eye must meet ALL ophthalmic inclusion and no exclusion criteria; Fellow Eye is the non-Study Eye. Fellow Eye may meet ophthalmic inclusion and exclusion criteria, but is not required.
  Eyes
    Open-angle glaucoma - Study Eye | 33 | 43 | 42 | 118
    Ocular hypertension - Study Eye | 32 | 22 | 22 | 76
    Open-angle glaucoma - Fellow Eye | 33 | 42 | 42 | 117
    Ocular hypertension - Fellow Eye | 32 | 23 | 22 | 77
Randomization Intraocular Pressure (Study Eye) [Count of Participants; unit: Participants] — Only the Study Eye of the 65 participants was measured in this table
  Participants
    Diurnal Mean < 26 mmHg | 49 | 49 | 48 | 146
    Diurnal Mean >=26 mmHg | 16 | 16 | 16 | 48
Study Eye Screening Corneal Thickness (micrometers) [Mean (Standard Deviation); unit: micrometer] — Only the Study Eye of the 65 participants was measured in this table
  micrometer | 544.8 (30.27) | 554.0 (28.57) | 554.7 (30.58) | 551.2 (30.00)
Study Eye Screening Intraocular Pressure (mmHg) [Mean (Standard Deviation); unit: mmHg] — Only the Study Eye of the 65 participants was measured in this table
  mmHg | 20.34 (1.981) | 20.54 (2.283) | 20.11 (2.003) | 20.33 (2.091)
Study Eye Baseline Diurnal Mean Intraocular Pressure (mmHg) [Mean (Standard Deviation); unit: mmHg] — Only the Study Eye of the 65 participants was measured in this table
  mmHg | 24.83 (1.559) | 25.16 (2.039) | 25.11 (1.967) | 25.03 (1.862)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Intraocular Pressure at Day 28 (Study Eye)
Description: Change from Baseline in Diurnal Mean IOP (mmHg) at Day 28 in the Study Eye -- ITT Population
Time Frame: Baseline to Day 28
Population: The ITT population will include all randomized subjects who have received at least one dose of study medication. This population will be the primary population for efficacy analyses and will be used to summarize all efficacy variables and will summarize subjects as randomized.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Groups:
- AKB-9778 4% QD + Latanoprost: • AKB-9778 4% QD (AM) and placebo for AKB-9778 4% ophthalmic solution daily (PM) plus latanoprost daily (PM) for 28 days
  Latanoprost ophthalmic solution: Latanoprost opthalmic solution to be dosed once daily
  razuprotafib: razuprotafib opthalmic solution
Arm/Group | AKB-9778 4% QD + Latanoprost | AKB-9778 4% BID + Latanoprost | Placebo Twice Daily + Latanoprost
Number analyzed (Participants) | 65 | 65 | 64
mmHg | -6.95 (0.258) | -7.95 (0.257) | -7.04 (0.259)
Statistical Analysis 1: Comparison: AKB-9778 4% QD + Latanoprost; Test type: Superiority; p = 0.8070, ANCOVA; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-0.63 to 0.81], Standard Error of Mean 0.366
Statistical Analysis 2: Comparison: AKB-9778 4% BID + Latanoprost; Test type: Superiority; p = 0.0130, ANCOVA; Mean Difference (Final Values) = -0.92, 95% CI 2-sided [-1.64 to -0.20], Standard Error of Mean 0.365

2. Secondary Outcome: Mean Change From Baseline in Diurnal Mean IOP at the Day 14 Visit (Study Eye)
Description: Change from Baseline in Diurnal Mean IOP (mmHg) at Day 14 in the Study Eye -- ITT Population
Time Frame: Baseline to Day 14
Population: The Intent-to-Treat population includes all randomized subjects who received at least one dose of study medication. the primary population for efficacy analyses and was used to summarize all efficacy variables and summarizes subjects as randomized.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | AKB-9778 4% QD + Latanoprost | AKB-9778 4% BID + Latanoprost | Placebo Twice Daily + Latanoprost
Number analyzed (Participants) | 65 | 65 | 64
mmHg | -6.75 (0.259) | -7.62 (0.258) | -7.03 (0.260)

3. Secondary Outcome: Mean Change From Baseline in Diurnal Mean IOP on Days 14 and 28 (Both Eyes)
Description: Mean change from baseline in diurnal mean IOP (measured in mmHg) at Day 14 and 28 in both eyes - ITT Population
Time Frame: Baseline to Day 14 and Baseline to Day 28
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | AKB-9778 4% QD + Latanoprost | AKB-9778 4% BID + Latanoprost | Placebo Twice Daily + Latanoprost
Number analyzed (Participants) | 65 | 65 | 64
Number analyzed (eyes) | 130 | 130 | 128
mmHg
  Baseline to Day 14 | -6.68 (0.250) | -7.53 (0.250) | -6.91 (0.252)
  Baseline to Day 28 | -6.83 (0.255) | -7.86 (0.255) | -6.93 (0.257)

4. Secondary Outcome: Observed Mean Diurnal Mean IOP on Days 14 and 28 (Both Eyes)
Description: Mean of the Diurnal Mean IOP (mmHg) at Day 14 and Day 28 in both eyes -- ITT Population
Time Frame: Baseline to Day 14 and Baseline to Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | AKB-9778 4% QD + Latanoprost | AKB-9778 4% BID + Latanoprost | Placebo Twice Daily + Latanoprost
Number analyzed (Participants) | 65 | 65 | 64
Number analyzed (eyes) | 130 | 130 | 128
mmHg
  Baseline to Day 14 | 18.01 (2.445) | 17.37 (2.272) | 17.95 (2.383)
  Baseline to Day 28 | 17.86 (2.514) | 17.03 (2.019) | 17.92 (2.580)

5. Secondary Outcome: Mean Observed IOP at Each Time Point on Days 14 and 28
Description: Mean observed IOP measured in mmHg at each time point on Days 14 and 28 (study eye) - ITT Population
Time Frame: Baseline to each timepoint on Day 14 and Baseline to each timepoint on Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AKB-9778 4% QD + Latanoprost | AKB-9778 4% BID + Latanoprost | Placebo Twice Daily + Latanoprost
Number analyzed (Participants) | 65 | 65 | 64
mmHg
  Day 14, 08:00 | 19.54 (2.970) | 18.25 (2.652) | 18.75 (3.289)
  Day 14, 10:00 | 17.98 (2.907) | 17.32 (2.772) | 18.02 (2.973)
  Day 14, 12:00 | 17.50 (3.059) | 17.25 (2.767) | 17.87 (2.624)
  Day 14, 16:00 | 17.52 (2.805) | 17.17 (2.762) | 17.56 (2.696)
  Day 28, 08:00 | 18.81 (2.977) | 18.13 (2.417) | 18.95 (2.986)
  Day 28, 10:00 | 17.97 (2.878) | 17.02 (2.558) | 17.90 (2.986)
  Day 28, 12:00 | 17.60 (2.791) | 16.55 (2.695) | 17.51 (2.914)
  Day 28, 16:00 | 17.35 (2.507) | 16.97 (2.377) | 17.82 (3.052)

6. Secondary Outcome: Mean Change From Baseline IOP at Each Time Point on Days 14 and 28
Description: Change from Baseline in Mean IOP (mmHg) at Each Time Point on Day 14 and Day 28 in the Study Eyes -- ITT Population
Time Frame: Baseline to each timepoint on Day 14 and Baseline to each timepoint on Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AKB-9778 4% QD + Latanoprost | AKB-9778 4% BID + Latanoprost | Placebo Twice Daily + Latanoprost
Number analyzed (Participants) | 65 | 65 | 64
mmHg
  Day 14, 08:00 | -6.66 (2.551) | -8.13 (3.225) | -7.59 (3.130)
  Day 14, 10:00 | -7.02 (2.607) | -7.88 (2.831) | -7.45 (2.388)
  Day 14, 12:00 | -6.79 (2.378) | -7.52 (2.761) | -6.83 (2.381)
  Day 14, 16:00 | -6.29 (2.698) | -7.10 (2.841) | -6.36 (2.332)
  Day 28, 08:00 | -7.39 (2.977) | -8.25 (2.826) | -7.38 (2.715)
  Day 28, 10:00 | -7.03 (2.665) | -8.19 (2.536) | -7.57 (2.549)
  Day 28, 12:00 | -6.69 (2.383) | -8.21 (2.486) | -7.18 (2.598)
  Day 28, 16:00 | -6.45 (2.279) | -7.30 (2.731) | -6.10 (2.593)

7. Secondary Outcome: Mean Percent Change From Diurnally Adjusted Baseline IOP at Each Time Point on Days 14 and 28
Description: Percent Change from Baseline IOP (mmHg) at Each Time Point on Day 14 and Day 28 in the Study Eyes -- ITT Population
Time Frame: Baseline to each timepoint on Day 14 and Baseline to each timepoint on Day 28
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | AKB-9778 4% QD + Latanoprost | AKB-9778 4% BID + Latanoprost | Placebo Twice Daily + Latanoprost
Number analyzed (Participants) | 65 | 65 | 64
percent change
  Day 14, 08:00 | -25.52 (1.292) | -30.41 (1.291) | -28.68 (1.301)
  Day 14, 10:00 | -28.09 (1.221) | -31.10 (1.219) | -29.29 (1.231)
  Day 14, 12:00 | -28.21 (1.213) | -30.19 (1.211) | -27.53 (1.219)
  Day 14, 16:00 | -26.48 (1.285) | -28.94 (1.287) | -26.61 (1.293)
  Day 28, 08:00 | -28.19 (1.218) | -30.96 (1.218) | -27.93 (1.227)
  Day 28, 10:00 | -28.12 (1.207) | -32.36 (1.205) | -29.70 (1.217)
  Day 28, 12:00 | -27.65 (1.209) | -33.09 (1.206) | -29.03 (1.215)
  Day 28, 16:00 | -27.21 (1.227) | -29.65 (1.229) | -25.58 (1.235)

8. Secondary Outcome: Mean Percent Change From Baseline in Diurnal Mean IOP on Days 14 and 28
Description: Percent Change from Baseline in Diurnal Mean IOP (mmHg) at Day 14 and Day 28 in the Study Eye -- ITT Population
Time Frame: Baseline to Day 14 and Baseline to Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | AKB-9778 4% QD + Latanoprost | AKB-9778 4% BID + Latanoprost | Placebo Twice Daily + Latanoprost
Number analyzed (Participants) | 65 | 65 | 64
percent change
  Baseline to Day 14 | -27.08 (7.875) | -30.29 (8.550) | -28.16 (7.931)
  Baseline to Day 28 | -27.83 (8.711) | -31.67 (7.219) | -28.19 (8.523)

9. Secondary Outcome: Percentages of Subjects Achieving Pre-Specified Mean, Mean Change, and Percent Mean Change in Diurnal Mean IOP Levels
Description: Percentages of Subjects Achieving Pre-Specified Mean, Mean Change, and Percent Mean Change in Diurnal Mean IOP Levels in Study Eye -- ITT Population
Time Frame: Baseline to Day 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AKB-9778 4% QD + Latanoprost | AKB-9778 4% BID + Latanoprost | Placebo Twice Daily + Latanoprost
Number analyzed (Participants) | 65 | 65 | 64
Participants
  Percentage of Subjects Achieving Pre-Specified Mean IOP: <=22 mmHg | 60 | 63 | 58
  Percentage of Subjects Achieving Pre-Specified Mean IOP: <=20 mmHg | 56 | 60 | 51
  Percentage of Subjects Achieving Pre-Specified Mean IOP: <=18 mmHg | 35 | 46 | 35
  Percentage of Subjects Achieving Pre-Specified Mean IOP: <=16 mmHg | 14 | 20 | 13
  Percentage of Subjects Achieving Pre-Specified Mean IOP : <=14 mmHg | 3 | 6 | 4
  Percentages of Subjects Achieving Mean Change (IOP Reduction from Baseline) : >=2 mmHg | 63 | 65 | 64
  Percentages of Subjects Achieving Mean Change (IOP Reduction from Baseline) : >=3 mmHg | 62 | 65 | 63
  Percentages of Subjects Achieving Mean Change (IOP Reduction from Baseline) : >=4 mmHg | 61 | 64 | 60
  Percentages of Subjects Achieving Mean Change (IOP Reduction from Baseline) : >=6 mmHg | 47 | 57 | 44
  Percentages of Subjects Achieving Mean Change (IOP Reduction from Baseline) : >=8 mmHg | 21 | 32 | 20
  Percentages of Subjects Achieving Mean Change (IOP Reduction from Baseline) : >=10 mmHg | 3 | 9 | 4
  Percent Mean Change in Diurnal Mean IOP Levels (IOP Percent Reduction from Baseline): >=5% | 63 | 65 | 64
  Percent Mean Change in Diurnal Mean IOP Levels (IOP Percent Reduction from Baseline): >=10% | 62 | 65 | 63
  Percent Mean Change in Diurnal Mean IOP Levels (IOP Percent Reduction from Baseline): >=15% | 61 | 64 | 59
  Percent Mean Change in Diurnal Mean IOP Levels (IOP Percent Reduction from Baseline): >=20% | 57 | 62 | 53
  Percent Mean Change in Diurnal Mean IOP Levels (IOP Percent Reduction from Baseline): >=25% | 43 | 55 | 41
  Percent Mean Change in Diurnal Mean IOP Levels (IOP Percent Reduction from Baseline): >=30% | 25 | 40 | 27
  Percent Mean Change in Diurnal Mean IOP Levels (IOP Percent Reduction from Baseline): >=35% | 13 | 18 | 11
  Percent Mean Change in Diurnal Mean IOP Levels (IOP Percent Reduction from Baseline): >=40% | 4 | 10 | 4

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected for the entire duration of the study, which was approximately 11 weeks.
Description: The Investigator is to report all directly observed AEs and all AEs spontaneously reported by the study subject. In addition, each study subject will be questioned about AEs at each visit following the initiation of treatment.
Arm/Group | AKB-9778 4% QD + Latanoprost | AKB-9778 4% BID + Latanoprost | Placebo BID + Latanoprost
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/65 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/65 | 0/64
Other Adverse Events (participants affected / at risk) | 30/65 | 43/65 | 19/64
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AKB-9778 4% QD + Latanoprost (N=65) | AKB-9778 4% BID + Latanoprost (N=65) | Placebo BID + Latanoprost (N=64)
Conjunctival hyperaemia (Eye disorders) | 26 (40) | 39 (63) | 9 (11) — ocular TEAE
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1) | 0 (0) — ocular TEAE
Dry Eye (Eye disorders) | 0 (0) | 1 (1) | 2 (2) — ocular TEAE
Eye Pruritus (Eye disorders) | 1 (1) | 2 (2) | 3 (3) — ocular TEAE
Eyelid margin crusting (Eye disorders) | 2 (2) | 1 (1) | 0 (0) — ocular TEAE
Iritis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) — ocular TEAE
Photophobia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) — ocular TEAE
Punctate keratitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) — ocular TEAE
Retinal artery emoblism (Eye disorders) | 1 (1) | 0 (0) | 0 (0) — ocular TEAE
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 1 (1) — ocular TEAE
Visual impairment (Eye disorders) | 1 (1) | 0 (0) | 0 (0) — ocular TEAE
Vitreous disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0) — ocular TEAE
Instillation site foreign body sensation (General disorders) | 0 (0) | 1 (1) | 0 (0) — ocular TEAE
Instillation site pain (General disorders) | 0 (0) | 2 (2) | 4 (4) — ocular TEAE
Instillation site pruritis (General disorders) | 0 (0) | 2 (2) | 0 (0) — ocular TEAE
Sensation of foreign body (General disorders) | 0 (0) | 1 (1) | 0 (0) — ocular TEAE
Migraine with aura (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) — ocular TEAE
Glossodynia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — non-ocular TEAE
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) — non-ocular TEAE
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — non-ocular TEAE
Dysgeusia (Nervous system disorders) | 3 (3) | 8 (8) | 1 (1) — non-ocular TEAE
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) — non-ocular TEAE

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Product acquired from Aerpio with limited transfer of documents. Site CTAs not provided.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-18): https://cdn.clinicaltrials.gov/large-docs/45/NCT04405245/Prot_SAP_000.pdf